CLINICAL TRIAL: NCT06606015
Title: Noninvasive Hemodynamics Assessment of Preterm Newborns With Successful Medical Closure of Patent Ductus Arteriosus
Brief Title: Noninvasive Hemodynamics Assessment of Preterms With Successful Medical Closure of PDA
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Lamiaa Khaled Zidan, Lecturer of Pediatrics, Tanta University
Other Study IDs: Hemodynamics with PDA closure
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Patent Ductus Arteriosus in Preterm Infants
Keywords: PDA; Electrical Cardiometry; hemodynamics
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Responders group:: included 26 preterm infants who successfully responded to medical PDA closure
  Interventions: Drug: I.V Paracetamol.; Device: Echocardiography.; Device: Electrical Cardiometry
- Non responders group:: included 17 preterm infants who didn't respond to medical PDA closure
  Interventions: Drug: I.V Paracetamol.; Device: Echocardiography.; Device: Electrical Cardiometry

INTERVENTIONS:
Drug: I.V Paracetamol. — Pharmacological thereby for hsPDA closure in the preterm neonates.
Device: Echocardiography. — It is routinely performed in neonates for PDA screening and detection of any other cardiac anomalies.
Device: Electrical Cardiometry — Non invasive hemodynamics monitoring

SUMMARY:
The aim of our study was to use Electrical Cardiometry EC to monitor hemodynamic alternations during pharmacological closure of hemodynamically significant patent ductus arteriosus (hsPDA) in preterm neonates

DETAILED DESCRIPTION:
PDA in the first three days of life is a normal physiologic remnant in healthy term neonates. Conversely, a PDA in preterm neonates causes significant clinical sequelae as a result from left to right shunting. It is widely recognized that a hemodynamically significant PDA is known to contribute to increased morbidity and mortality. The increase in pulmonary blood flow in the setting of prematurity leads to pulmonary edema, noncompliant lungs, and worsening of respiratory status. Other sequelae of a hemodynamically significant PDA include intraventricular hemorrhage, necrotizing enterocolitis, congestive heart failure, and failure to thrive.

Echocardiography is often used to evaluate hemodynamic significance of PDA. In general, pharmacological closure of PDA is less successful in infants with ductal diameter >2mm. Lower ductal maximum velocity, which is usually associated with a larger PDA or higher pulmonary pressure, is another predictor of treatment failure .

The use of echocardiography to gather meaningful hemodynamic data often necessitates serial assessments that can be tedious and labor-intensive. Electrical cardiometry (EC) is a non-invasive, impedance-based monitor that provides absolute cardiac output estimates in clinical practice. Unlike echocardiography, EC is simple to apply, continuous in measurements and not operator dependent.

ELIGIBILITY:
Inclusion Criteria:

* All preterm newborns who were admitted throughout the duration of the research.

Exclusion Criteria:

* Newborn with congenital heart diseases.
* Newborn with acquired heart diseases (viral myocarditis)
* Newborn with dysrhythmias
* Newborn with symptomatic cardiac dysfunction secondary to extra cardiac diseases
* Newborn with significant pulmonary hypertension or systemic hypertension

Ages: 24 Hours to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study included 43 preterm neonates with hemodynamically significant PDA who received IV paracetamol as PDA medical closure. They were subdivided into 2 main groups responders and non responders to the PDA closure treatment.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Stroke volume (SV) | 6 months
  Electrical cardiometry provides non-invasive hemodynamic monitoring. Electrical cardiometry provided a tool for continuous and non-invasive monitoring of Preterm Newborns with successful medical closure of PDA by evaluating: Stroke volume (SV): higher in non-responders.
Cardiac output (CO) | 6 months
  Electrical cardiometry provides non-invasive hemodynamic monitoring. Electrical cardiometry provided a tool for continuous and non-invasive monitoring of Preterm Newborns with successful medical closure of PDA by evaluating: Cardiac output (CO): higher in non-responders.
Systemic vascular resistance (SVR) | 6 months
  Electrical cardiometry provides non-invasive hemodynamic monitoring. Electrical cardiometry provided a tool for continuous and non-invasive monitoring of Preterm Newborns with successful medical closure of PDA by evaluating:
  Systemic vascular resistance (SVR): higher in responders.
Total fluid content (TFC) | 6 months
  Electrical cardiometry provides non-invasive hemodynamic monitoring. Electrical cardiometry provided a tool for continuous and non-invasive monitoring of Preterm Newborns with successful medical closure of PDA by evaluating:
  3. Total fluid content (TFC): higher in non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Elmahdy, Professor of Pediatrics, Study Director — Tanta University
Locations (1):
- Faculty of Medicine, Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided